CLINICAL TRIAL: NCT05453708
Title: Maternal Risk Factors for Autism Spectrum Disorders: A Case-Control Approach
Status: Completed | Type: Observational
Sponsor: Walden University (Other)
Responsible Party: Principal Investigator, Michael Haniff, Principal Investigator, Walden University
Other Study IDs: 06-16-22-0412467
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Autism; Autism Spectrum Disorder; Autistic Disorder; Pregnancy Related; Diet, Healthy; Diet; Deficiency; Folate Deficiency; Folic Acid Deficiency; Folic Acid Overdose
Keywords: Diet; Maternal diet; Autism pregnancy; Perinatal; Folate; Folic Acid
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Malnutrition; Folic Acid Deficiency | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Risk: Survey for mothers 18 years or older with a child aged 3-12 years who has an official ASD diagnosis from a clinician.
  Interventions: Other: Survey
- Controls: Survey for mothers 18 years or older of children aged 3-12 years who do not have an ASD diagnosis so comparisons can be made between groups.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — One 15-20-minute survey

SUMMARY:
New research suggests that about 1 in 8 children may be diagnosed with an autism spectrum disorder (ASD) in the United States. This could be due to several reasons which remain unknown. This study invites mothers who have given birth to children in the United States to share their experiences with diet and supplementation during pregnancy. The purpose of this study is to understand the role of a mother's diet, social standing, and supplementation with folate or folic acid may have on her child's future development of autism. Comparisons will be made between mothers of children who have a child with an official ASD diagnosis from a clinician to mothers of children without an ASD diagnosis. Findings from this study can be used to help identify risk factors for ASD risk.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) are a broad range of conditions characterized by social skills, repetitive behaviors, speech, and nonverbal communication challenges. Current prevalence estimates assert that 2.3% of children aged eight years or older live with an ASD, an increase from 1.5% in 2012. Estimates suggest that 1 in 44 children will be diagnosed with ASD. A child diagnosed on the spectrum faces several challenges and may require support from a caregiver, possibly across the lifespan. ASD etiology remains elusive, but research suggests there may be a link to genetic, environmental, and dietary risk factors while in-utero.

Further evidence suggests a folate/folic acid link during the peri-conceptual period. Prior folate/folic acid studies suggest a U-shaped relationship between maternal multivitamin supplementation. High maternal plasma folate and B12 levels are associated with the risk of ASD.

This study aims to apply a case-control approach to understand the role of folate/folic over- or under-supplementation, maternal sociodemographics, and diet during pregnancy on ASD risk.

ELIGIBILITY:
Inclusion Criteria:

* Mothers 18 years or older with a child aged 3-12 years who have an official ASD diagnosis from a clinician
* Mothers 18 years or older of children aged 3-12 years who do not have an ASD diagnosis so comparisons can be made between groups

Exclusion Criteria:

* Mothers outside of the United States
* Mothers less than 18 years of age
* Mothers who have not given birth to their child or who used a surrogate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This survey asks mothers to provide information about their experiences with diet and supplementation during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Association between maternal folate intake during pregnancy and the occurrence of ASD in the offspring via questionnaire. | 42 weeks gestation
  Number of participants with a child diagnosed with ASD who used multivitamins or folate/folic acid supplements during pregnancy as assessed by the questionnaire.

SECONDARY OUTCOMES:
Association between mother's co-morbidities and the occurrence of ASD in offspring via questionnaire. | 42 weeks gestation
  Number of participants with a child diagnosed with ASD who also have a comorbidity or developed a comorbidity during pregnancy as assessed by the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Haniff, Principal Investigator — Student
Locations (1):
- Walden University, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No